CLINICAL TRIAL: NCT07203599
Title: A Randomized Controlled Clinical Study on the Treatment of Androgenetic Alopecia in Young Men With Umbilical Cord Mesenchymal Stem Cell Exosomes
Brief Title: A Study on the Treatment of Androgenetic Alopecia in Young Men With Umbilical Cord Mesenchymal Stem Cell Exosomes
Acronym: MSCs treatment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LL-KY-2024218-04
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Androgenic Alopecia
Keywords: androgenic alopecia; human umbilical cord mesenchymal stem cell exosomes
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): Participants will receive one injection site for each 1 cm² of hair loss area, delivering a dosage of 1.0×10^8 particles of hUCMSC-sEV per site.
  Interventions: Drug: Human umbilical cord mesenchymal stem cell exosomes
- Group B (Experimental): Participants will receive one injection site for each 1 cm² of hair loss area, delivering a dosage of 1.0×10^9 particles of hUCMSC-sEV per site.
  Interventions: Drug: Human umbilical cord mesenchymal stem cell exosomes
- Group C (Experimental): Participants will receive one injection site for each 1 cm² of hair loss area, delivering a dosage of 1.0×10^10 particles of hUCMSC-sEV per site.
  Interventions: Drug: Human umbilical cord mesenchymal stem cell exosomes
- hUCMSC-sEV treatment group (Experimental): Participants will receive one injection site for each 1 cm² of hair loss area with the optimal dose of hUCMSC-sEV.
  Interventions: Drug: Human umbilical cord mesenchymal stem cell exosomes
- Minoxidil treatment group (Active Comparator): Participants will get 1 mL of minoxidil administered daily to the area of hair loss.
  Interventions: Drug: Minoxidil 5% Topical Solution

INTERVENTIONS:
Drug: Human umbilical cord mesenchymal stem cell exosomes — Human umbilical cord mesenchymal stem cell exosomes are nanoscale vesicles released by mesenchymal stem cells from the umbilical cord. These exosomes act as natural carriers, transferring proteins, microRNAs (miRNAs), and other molecules to recipient cells. This communication helps the exosomes exert therapeutic effects, promoting tissue repair, reducing inflammation, and mediating cell-to-cell interactions in various disease models.
  Other Names: hUCMSC-sEV
  Arms: Group A; Group B; Group C; hUCMSC-sEV treatment group
Drug: Minoxidil 5% Topical Solution — Topical minoxidil is a medicine used to help regrow the hair on your scalp. It works by increasing the blood flow to your hair and helps stimulate your hair follicles to grow.
  Arms: Minoxidil treatment group

SUMMARY:
This clinical trial aims to determine the efficacy of human umbilical cord mesenchymal stem cell exosomes (hUCMSC-sEV) in treating androgenic alopecia in young men. It will also investigate the safety of hUCMSC-sEV. The primary inquiry it seeks to address is:

* Do hUCMSC-sEV demonstrate efficacy in the treatment of androgenic alopecia in young men?
* Do hUCMSC-sEV safely used to treat androgenic alopecia in young men?

The clinical trial has two parts. The Phase I study is a dose-escalation trial. Researchers will determine the appropriate dosage of hUCMSC-sEV. The Phase II study is a randomized controlled trial. Researchers will evaluate hUCMSC-sEV against a placebo (minoxidil tincture) to determine the efficacy of hUCMSC-sEV in treating androgenic alopecia in young men.

In the phase I study, participants will be categorized into three dosage groups: A, B, and C. In Group A, one injection site will be allocated for each 1 cm² of hair loss area, delivering a dosage of 1.0×10^8 particles per site. In Group B, the dosage will be 1.0×10^9 particles per site. In Group C, the dosage will be 1.0×10^10 particles per site. Participants will attend the clinic at weeks 0, 2, 4, and 6 for treatment and assessments. Participants will also attend the clinic for follow-up examinations at weeks 8, 12, and 24.

In the phase II study, participants will be randomly allocated in a 1:1 ratio to two groups: the hUCMSC-sEV treatment group and the minoxidil treatment group. hUCMSC-sEV treatment group: the appropriate dose of hUCMSC-sEV for the phase II study was determined based on assessments of safety, tolerability, and preliminary efficacy from the phase I study. Participants will receive one injection site for each 1 cm² of hair loss area. Participants will attend the clinic for therapy and assessments at weeks 0, 2, 4, and 6. Minoxidil treatment group: participants will get 1 mL of minoxidil administered daily to the area of hair loss for 12 consecutive weeks. All patients will attend the clinic for follow-up examinations at weeks 8, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male patients aged 18-35 2. Clinically diagnosed with androgenic alopecia, Hamilton Norwood Scale III-V 3. Patients who voluntarily participate in clinical trials and sign informed consent forms

Exclusion Criteria:

* 1. Known alcohol allergy 2. Patients with severe primary diseases of cardiovascular, cerebrovascular, liver, kidney, endocrine, or hematopoietic system 3. Patients with other scalp diseases or hair loss diseases 4. Patients with severe mental illness and cognitive impairment 5. Patients with poor nutritional status and low immune function 6. Within 1 year, those who have used systemic corticosteroids, immunosuppressants, cytotoxic drugs, and peripheral vasodilators 7. Within 6 months, those who have used systemic or local drugs to treat hair loss, such as finasteride, minoxidil, etc 8. Within 3 months, those who have received other clinical trial drugs 9. Family genetic history or other criteria considered unsuitable by researchers

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Hair density | From the first treatment to 24 weeks.
  Hair density will be measured by dermoscopy at weeks 0, 8, 12 and 24.
Hair diameter | From the first treatment to 24 weeks.
  Hair diameter will be measured by dermoscopy at weeks 0, 8, 12 and 24.
Hair count | From the first treatment to 24 weeks.
  Hair count will be measured by dermoscopy at weeks 0, 8, 12 and 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No